CLINICAL TRIAL: NCT03985696
Title: Exosomes and Resistance to Immunotherapy in Aggressive Non-Hodgkin B-cell Lymphomas (B-NHL)
Brief Title: Exosomes and Immunotherapy in Non-Hodgkin B-cell Lymphomas
Acronym: ExoReBLy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 87RI18_0025 (ExoReBLy)
Record Dates: First submitted 2019-06-11; First posted 2019-06-14 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Lymphoma, B-cell, Aggressive Non-Hodgkin (B-NHL)
Keywords: B cells; exosomes; immunotherapy; Lymphomas; DLBCL
MeSH Terms: conditions — Lymphoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with DLBCL (Experimental)
  Interventions: Other: blood sample
- Healthy volunteers (Active Comparator)
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample — 1 blood volume (5-7 ml EDTA)

SUMMARY:
Diffuse large B-cell lymphomas (DLBCL) are highly aggressive and heterogeneous B-cell lymphoma that would imminently be fatal without treatment. Monoclonal anti-CD20 antibody, rituximab, in combination of CHOP chemotherapy (R-CHOP) is widely used with favourable results. Although more than half of patients achieve long-term remission, many are not cured with this immunotherapy. Suboptimal response and/or resistance to rituximab have remained a challenge in the therapy of DLBCL but also of all B-NHL. Exosomes are microvesicles released from tumor B cells that are found in plasma of patients with B-NHL. Exosomes carry therapeutic targets (as CD20, PDL-1) and could act as "decoy-receptors" for immunotherapy. Our objective is to precise, in aggressive B-NHL, the role of exosomes in immunotherapy escape.

DETAILED DESCRIPTION:
Diffuse large B-cell lymphomas (DLBCL) are highly aggressive and heterogeneous B-cell lymphoma that would imminently be fatal without treatment. Monoclonal anti-CD20 antibody, rituximab, in combination of CHOP chemotherapy (R-CHOP) is widely used with favourable results. Although more than half of patients achieve long-term remission, many are not cured with this immunotherapy. Decreased CD20 expression has been postulated to be one of the most important contributing to rituximab resistance. Moreover, R-CHOP therapies are sometimes ineffective, and new treatment strategies based notably on host immune responses modulation are being explored. Among them, programmed cell death ligand 1 (PD-L1) protein was identified as a potent predicting biomarker in DLBCL. Exosomes are small membrane vesicles secreted by several cell types during exocytic fusion of multivesicular bodies with the plasma membrane. Many cancer cells have been shown to secrete exosomes in greater amounts than normal cells. Exosome secretion may contribute to drug resistance. Indeed, exosome release from B-cell Non-Hodgkin Lymphoma (B-NHL), by the expression of CD20, has been suggest to act as decoy targets upon rituximab exposure, allowing lymphoma cells to escape from humoral immunotherapy. Finally, as exosome composition seems to be cell and tissue specific, they are highly suitable to serve as diagnostic markers.

Our hypothesis is that high expression of the immunotherapeutic targets (CD20, PD-L1) on exosomes derived from aggressive or resistant B-NHL may allow tumor cells to escape therapeutic antibodies, and thus contribute in vivo to therapeutic resistance. For this objective, we will used exosomes derived from DLBCL human cells and exosomes isolated from plasma of DLBCL patients. We will analyze, on these microvesicles, CD20 and PDL-1 expression in function of DLBCL sub-types and outcome of patients. Moreover, exosome capacity to interfere with immunotherapy will be also studied from in vitro and in vivo (xenografts) models.

ELIGIBILITY:
Inclusion Criteria :

* patients over 18 years old with DLBCL at diagnostic or relapsed patients after R-CHOP therapy.
* Healthy volunteers over 18 years old

Exclusion Criteria:

* other B cell diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-07-02 (Actual); Primary Completion 2025-07-02 (Estimated); Study Completion 2025-07-02 (Estimated)

PRIMARY OUTCOMES:
Quantification of CD20 and PDL-1 in exosomes purified from cell cultures of DLBCL human cell lines and from Healthy volunteers | Month 36
  From D0 until the end of the inclusion period (36 months)

SECONDARY OUTCOMES:
Evaluation if peripheral exosomes can be used as novel diagnostic biomarkers in DLBCL | Month 36
  To analyze the prognostic value of exosomal markers on therapeutic response and patient outcome, each patient included in the study at diagnostic (D0) will be followed up until 36 months after inclusion.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Limoges, Limoges, France

IPD SHARING:
Plan to Share IPD: No